CLINICAL TRIAL: NCT04188015
Title: A Phase 1b, Randomized, Double-masked, Sham-controlled Study of ANX007 Administered as Intravitreal Injections to Assess Safety and Tolerability in Participants With Primary Open-angle Glaucoma
Brief Title: Study of ANX007 in Participants With Primary Open-angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANX007-GLA-02
Record Dates: First submitted 2018-12-13; First posted 2019-12-05 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2.5mg ANX007 (Experimental): 1 in every 3 subjects will be randomized to 2.5mg dose of ANX007.
  Interventions: Biological: 2.5mg ANX007
- 5.0mg ANX007 (Experimental): 1 in every 3 subjects will be randomized to 5.0mg dose of ANX007.
  Interventions: Biological: 5.0mg ANX007
- Sham Procedure (Sham Comparator): 1 in every 3 subjects will have a sham procedure performed instead of receiving ANX007.
  Interventions: Other: Sham Procedure

INTERVENTIONS:
Biological: 2.5mg ANX007 — A single dose of 2.5mg ANX007 will be administered via IVT injection into the study eye at Day 1 and Day 29.
  Arms: 2.5mg ANX007
Biological: 5.0mg ANX007 — A single dose of 5.0mg ANX007 will be administered via IVT injection into the study eye at Day 1 and Day 29.
  Arms: 5.0mg ANX007
Other: Sham Procedure — The sham injection is preformed by applying pressure to the eye at the location of a typical IVT injection using the blunt end of a syringe without a needle.
  Arms: Sham Procedure

SUMMARY:
This is a double-masked, randomized, sham-controlled study evaluating two dose levels of ANX007 vs sham, administered as repeat Intravitreal (IVT) injections in patients with Primary Open-angle Glaucoma.

DETAILED DESCRIPTION:
This is a phase 1b, double-masked, sham-controlled study evaluating 2 dose levels of ANX007 administered as 2 IVT injections separated by 4 weeks. Approximately 15-29 subjects will be enrolled. An interim analysis of the initial set of 15 participants may be conducted. Based on this analysis, an additional 10-14 participants may be enrolled at a 1:1 ratio to receive one of the two dose levels.

The primary objective is to evaluate the safety and tolerability of repeat IVT injections of ANX007 in participants with primary open-angle glaucoma. Secondary objectives are to evaluate the anterior chamber fluid pharmacokinetics (PK) of ANX007, PD effect of ANX007 on anterior chamber fluid C1q activity, and immunogenicity. An exploratory objective will evaluate ocular PD effect of ANX007.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18 years, and above.
2. Diagnosis of primary open-angle glaucoma.
3. Ability to perform a reliable visual field test in the study eye with a cutoff of 33% for fixation losses and 33% for false-positive response rates.
4. Intraocular pressure (IOP) <21 mm Hg at screening and Day 1.
5. The IOP treatment regimen in the study eye should be stable for at least 4 weeks prior to injection, with no change in the IOP treatment regimen anticipated throughout study participation.
6. Ability to comply with the requirements of the study and complete the full sequence of protocol specified injections, procedures, and evaluations.

Exclusion Criteria:

1. Extensive glaucomatous visual-field damage with a mean deviation worse than -18 dB on Humphrey visual field testing.
2. Any current or prior ocular pathology, other than glaucoma, which could interfere with the conduct of the study including, but not limited to, retinal or optic nerve disease and media opacity in the study eye.
3. History of intraocular inflammatory or infectious eye disease in the study eye.
4. Ocular trauma in the study eye within the preceding 6 months.
5. A history of uncomplicated cataract surgery less than 3 months prior to injection, or trabeculectomy, iridotomy, or other ocular procedures in the study eye that could affect drug distribution and excretion.
6. Any abnormality preventing reliable tonometry in the study eye.
7. Concurrent use of glucocorticoid medications administered by any ocular or systemic route. Nasal, inhaled, and dermatologic (if not administered around the eyes) glucocorticoids are permitted.
8. Receiving monoamine oxidase inhibitor therapy or patient-reported hypersensitivity to any component of apraclonidine, brimonidine, clonidine, phenylephrine, povidone iodine, proparacaine, or ANX007.
9. Active or history of malignancy within the past 5 years with the exception of curatively treated, basal cell carcinoma.
10. Previous treatment with another humanized monoclonal antibody, Fab or Fab'2.
11. History of any autoimmune or neurologic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of ANX007 in participants with primary open-angle glaucoma as measured by occurrence of treatment-emergent adverse events. | Day 85

SECONDARY OUTCOMES:
Evaluate PK parameters of ANX007 in serum after repeat injections | Day 29
  Maximum Serum Concentration (Cmax) of ANX007
Evaluate PK parameters of ANX007 in serum after repeat injections | Day 29
  Area Under the Curve (AUC) of ANX007
Evaluate PK parameters of ANX007 in aqueous humor after repeat intravitreal injections | Day 29
  Maximum aqueous humor Concentration (Cmax) of ANX007
Evaluate PK parameters of ANX007 in aqueous humor after repeat intravitreal injections | Day 29
  Aqueous humor Area Under the Curve (AUC) of ANX007
Evaluate PD parameters of ANX007 in aqueous humor after repeat intravitreal injections | Day 29
  Maximum C1q concentration (Cmax) in aqueous humor
Evaluate PD parameters of ANX007 in aqueous humor after repeat intravitreal injections | Day 29
  C1q area under the curve (AUC) in aqueous humor
Evaluate PD parameters of ANX007 in serum after repeat intravitreal injections | Day 29
  Maximum C1q concentration (Cmax) in serum
Evaluate PD parameters of ANX007 in serum after repeat intravitreal injections | Day 29
  C1q concentration area under the curve (AUC) in serum
Immunogenicity of ANX007 as measured by serum anti-drug antibodies (ADA) after repeat intravitreal injections of ANX007 | Day 84
  Incidence of positive antibody titre against ANX007 in serum

CONTACTS AND LOCATIONS:
Overall Officials: Eric Humphriss, Study Director — Annexon Biosciences
Locations (2):
- United States (2):
  - Eye Research Foundation, Newport Beach, California
  - Stanford Health Care, Stanford, California

REFERENCES:
- See also: Related Info — http://www.annexonbio.com